CLINICAL TRIAL: NCT06135480
Title: Subcision With Platelet-Rich Plasma and Microneedling Versus Subcision With Saline and Micro-needling in Treatment of Posttraumatic Scars: Randomized Clinical Trial
Brief Title: Subcision With PRP and Microneedling Versus Subcision With Saline and Micro-needling in Treatment of Posttraumatic Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Howida Omar Twisy, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Post traumatic scars treatment
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Post-Traumatic Scar
MeSH Terms: interventions — Sodium Chloride; Percutaneous Collagen Induction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined subcision with platelet-rich plasma and microneedling group (Active Comparator)
  Interventions: Other: subcision ,PRP or saline and microneedling
- combined subcision with saline and microneedling group (Active Comparator)
  Interventions: Other: subcision ,PRP or saline and microneedling

INTERVENTIONS:
Other: subcision ,PRP or saline and microneedling — minimally invasive procedures

SUMMARY:
Compare different minimally invasive approaches to reach optimum improvement by comparing the efficacy and safety of both combined subcision with platelet-rich plasma and microneedling versus combined subcision with saline and microneedling in the treatment of post-traumatic scars.

DETAILED DESCRIPTION:
The scars at the level of the skin represent a normal and inevitable process of healing traumatic or surgical lesions, but except for the appearance of the skin, they also have a profound psychological impact . Thus, people with scars try to integrate them into their sense of self to gain psychological acceptance .

Many treatment options have been developed for the management of traumatic scars .Surgical intervention is an invasive technique, surgery has a high risk of inducing new scar formation .

Non-surgical approaches for the treatment of traumatic scars include topical treatments and minimally invasive approached as subcision,microneedling and laser.

Autologous platelet-rich plasma is plasma with a higher concentration of platelets than normally found, it can enhance wound healing which has been demonstrated in controlled studies for soft and hard tissues . The application of autologous platelet-rich plasma to surgical wounds has been shown to accelerate tissue repair and reduce postoperative pain .

Subcision is a procedure in which a needle is inserted under the skin and passed in multiple directions . Although subcision is adequate as a stand-alone treatment, improved results are achieved when it is combined with other modalities.

Microneedling is a percutaneous collagen induction therapy that causes skin resurfacing. It involves using fine needles to create controlled microdermal injuries starting a complex cascade of growth factors that end in collagen remodeling .

Because of the different treatment options available for this common problem, the current work aimed to combine and compare different minimally invasive approaches to reach optimum improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with posttraumatic scars
* Age more than 12 years

Exclusion Criteria:

* Patients with platelet or blood clotting disorders, and chronic liver or autoimmune diseases.
* Patients with chronic debilitating diseases, uncontrolled systemic infection, or keloid tendency or with unrealistic expectations.
* Pregnant females.
* Patients who did not complete the treatment sessions or the follow-up period.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Scar severity grading | after 1 month of treatment completion.
  Scar severity grading will be evaluated by blinded dermatologist

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Twisy HO. Subcision with platelet-rich plasma and microneedling versus subcision with saline and micro-needling in posttraumatic scars. Arch Dermatol Res. 2024 Aug 19;316(8):537. doi: 10.1007/s00403-024-03226-3. PMID 39158761